CLINICAL TRIAL: NCT04909060
Title: Does the Newborn Infant Parasympathetic Evaluation (NIPE) Index Predict Postsurgical Pain in Children
Acronym: NIPE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Responsible Party: Principal Investigator, Gianluca Bertolizio, MD, FRCPC, Associate Professor, Anesthesiologist, McGill University Health Centre/Research Institute of the McGill University Health Centre
Other Study IDs: Observational
Record Dates: First submitted 2021-05-26; First posted 2021-06-01 (Actual); Last update posted 2023-05-03 (Actual); Status verified 2023-05

CONDITIONS: Post Operative Pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Device: noninvasive blood pressure, 3 lead ECG, peripheral oxygen saturation — Children between 1 and 3 years old, scheduled for elective adeno-tonsillectomy, tonsillectomy or adenoidectomy and with no neurological or cardiac congenital deficits, no cardiac arrythmias (non-sinus rhythm), no implanted pacemakers, nor with a history of prolonged resuscitation at birth, and chronic therapy with drugs that have known effects on sympathetic and parasympathetic activity, ASA physical status III or higher and parent/guardian refusal will have a NIPE placed on their electrocardiogram, at least 20 minutes before the expected end of the surgery, the NIPE monitor will be connected to the anesthesia monitor at the end of the surgery, when the patient is considered ready to be transferred to the PACU, the NIPE will be disconnected and reconnected to the patient monitor once in PACU. Values will be recorded until the patient meets the discharge criteria from PACU not before 2hours

SUMMARY:
An investigation to find out if Newborn Infant Parasympathetic Evaluation (NIPE) index predicts postsurgical pain in children, since NIPE is thought to may be of guide to the appropriate therapy in a timely and objective manner, thereby improving patient safety, parental satisfaction, and reducing healthcare costs. We think that, validating the utility of NIPE in children under 3 years of age will allow the implementation of a novel pain assessment tool to our current practice of anesthetic care. This will improve the perioperative pain management, in particular for patients who are unable to communicate pain, with the potential to reduce detrimental consequences of postoperative pain.

And also determining the relationship between the NIPE scores and validated FLACC scale for post-operative pain and PAED scale during the recovery from anesthesia and also to determine whether NIPE values at extubation correlates with the incidence of moderate and/or severe pain in PACU.

DETAILED DESCRIPTION:
Pain represents a sensorial experience in response to tissue damage, that does not only affects the emotional and functional domains of an individual, but also leads to multiple detrimental, unanticipated and long-lasting consequences. In fact, pain has been associated with cognitive disturbances, increase in cancer recurrence, impairment in brain development and impairment of the immune system. Pain associated with surgical stress delays postoperative ambulation and discharge, promotes the development of chronic postoperative pain, and increases morbidity and mortality.

Despite the advancement in analgesics and pain control modalities, severe postoperative pain is present in up to 40% of patients. Improved pain management based on an accurate assessment of patients' pain intensity has been associated with better patient outcomes. As a consequence, standardized, validated instruments to facilitate pain evaluation have been recommended by the American Society of Anesthesiologists (ASA) Task Force on Acute Pain Management. Self-report scales, behavioral scales and physiological measures have been developed to assess pain after surgery. These tools, however, are applicable only in awake, cooperative patients and have limited value in uncooperative and non-verbal patients, such as young children.

In recent years, investigations have focused on parasympathetic tone activity as an indirect assessment of the level of pain. While heart rate variability (HRV) is affected by the balance between sympathetic and parasympathetic tone, the high frequency changes of HRV is primarily mediated by and specific to the parasympathetic nervous system. The phenomena of pain, fear, anxiety and intraoperative nociception have proven to be accompanied by changes in HRV. In pediatric patients, HRV analysis correlates with prolonged pain and newborn comfort.

The newborn infant parasympathetic evaluation (NIPE) is a non-invasive, standardized continuous measurement of HRV. The cardiac signal is extrapolated from the electrocardiogram and respiratory rate (RR) series are computed between two heart beats, resampled at 8 Hz, mean centered and normalized over a 64-second moving window. A wavelet based high pass filter over 0.15 Hz is applied in order to keep parasympathetic related variations only, which are mainly influenced by the respiratory cycle. The NIPE monitor displays two averaged measurements: the average NIPE (NIPEa) results from the average of NIPE measured over the previous 20 minutes, and current NIPE (NIPEc) results from the average of NIPE measured over the previous 64 seconds. A non-disclosed algorithm derived from the high frequency changes of the HRV calculates a score between 0 and 100, where a score of 0 indicates minimal parasympathetic tone and maximal nociception and a score of 100 indicates maximal parasympathetic tone and minimal nociception.

The NIPE index is a modification of Analgesia Nociception Index (ANI) and was developed for infants and young children who have higher baseline HR resulting in a lower possible variability. The ANI has shown a good performance in predicting intraoperative nociceptive stimuli in animals, adults7, and older children. In adults, ANI was able to predict the incidence of moderate/severe pain postoperatively and in critically ill patients.

To date, NIPE has shown promising results in the assessment of intraoperative and procedural pain, and neonatal comfort. On the contrary, there is a paucity of literature examining the usefulness of NIPE in guiding postoperative pain management in young children.

The current standard of care relies on scales incorporating various behavioural parameters to evaluate the likelihood of pain and the need for analgesic medication. The most commonly used scales in preschool children, who are not able to complete self-assessments, are the Children's Hospital of Eastern Ontario Pain Scale (CHEOPS), the Face, Legs, Activity, Cry and Consolability Scale (FLACC), and the Children and Infants' Postoperative Pain Scale (CHIPPS). These scales are limited in their dependence on examiner's ability to use the tool and training. Recently, the Pediatric Critical-Care Pain Observation Tool (P-CPOT) has been validated in critically ill children, but no data on postsurgical pediatric patients has been published.

The postoperative pain assessment in small children may be confused with Emergence Delirium (ED), an anesthesia related complication that affects 25% children undergoing surgery. ED is associated with significant adverse effects including injury to the patient and personnel, damage to incision sites, exacerbated parental anxiety, and increased nursing requirements, further resulting in an increased burden and cost to the healthcare system. Once ED occurs, extra nursing care may be necessary, as well as supplemental sedative and/or analgesic medications, which may delay patient discharge. Children showing ED after anaesthesia are seven times more likely to have new-onset separation anxiety, apathy, eating and sleeping problems. To date, only the Pediatric Anesthesia Emergence Delirium (PAED) scale has been validated in the pediatric population, but its capability to discriminate between ED and pain has been recently questioned.

In the absence of appropriate diagnostic tools, the management of pain or emergence delirium may be delayed while attempting to treat the other possible confounding conditions that may similarly occur in the Post Anesthesia Care Unit (PACU).

ELIGIBILITY:
Inclusion Criteria:

* Children between 3 and 7 years old, scheduled for elective adeno-tonsillectomy, tonsillectomy or adenoidectomy.
* Only patients whose parents are fluent in French or English will be enrolled

Exclusion Criteria:

* Patients with neurological or cardiac congenital deficits, with cardiac arrythmias (non-sinus rhythm)
* Implanted pacemakers, with a history of prolonged resuscitation at birth, on chronic therapy with drugs that have known effects on sympathetic and parasympathetic activity (antimuscarinics, beta 2 adrenergic agonists
* Alpha 1-adrenergic antagonists or antiarrhythmic agents,
* Tricyclic antidepressants.
* ASA physical status III or higher and parent/guardian refusal.
* Patients be scheduled for surgery without an appointment at the Montreal Children's Hospital (MCH) Preoperative Clinic
* A surgery appointment within 24 hours of surgery, will not be enrolled into the study.

As this study will be conducted with only one NIPE monitor, and it will be devoted to the patient for about 1.5 hours, two consecutive patients cannot be enrolled in the study. In this case, the second patient will be considered eligible but excluded, and data will not be collected.

Ages: 3 Years to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Preschool children
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2024-09 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Validation of NIPE as a tool to prevent and assess postoperative pain will improve monitoring of children and potentially their outcome | 24 Hours

CONTACTS AND LOCATIONS:
Locations (1):
- Montreal Children's Hospital, Montreal, Quebec, Canada

REFERENCES:
- [Derived] Chisling S, Jette E, Engelhardt T, Ingelmo P, Poulin-Harnois C, Garbin M, Wasserman S, Bertolizio G. Does heart rate variability using the Newborn Infant Parasympathetic Evaluation index identify postsurgical pain levels and emergence delirium in toddlers? A prospective observational study. Can J Anaesth. 2024 Aug;71(8):1117-1125. doi: 10.1007/s12630-024-02764-8. Epub 2024 May 8. PMID 38720113